CLINICAL TRIAL: NCT00703924
Title: Topical Treatment of Cutaneous Leishmaniasis With WR 279,396: a Phase 2 Study in the Old World
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A-9768.1; IND 50098 (Other: FDA)
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Cutaneous Leishmaniasis
Keywords: cutaneous leishmaniasis topical treatment safety efficacy
MeSH Terms: conditions — Leishmaniasis, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- WR 279,396 (Experimental): WR 279,396 is a topical antibiotic cream containing paromomycin and gentamicin
  Interventions: Drug: WR 279,396
- Placebo (Placebo Comparator): Topical cream vehicle containing all of the components in WR 279,396 except the active ingredients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WR 279,396 — A topical cream containing 15% paromomycin and 0.5% gentamicin. Approximately 0.0005 mL per mm2 of skin lesion
  Other Names: Paromomycin topical cream
  Arms: WR 279,396
Drug: Placebo — Topical cream vehicle. Approximately 0.0005 mL per mm2 of skin lesion
  Other Names: Topical vehicle placebo
  Arms: Placebo

SUMMARY:
This study is to determine the effectiveness and safety of WR 279,396, a topical cream for the treatment of cutaneous leishmaniasis. This study is to be conducted with a placebo control under double-blind conditions in a local population group in Tunisia where leishmaniasis is endemic.

DETAILED DESCRIPTION:
WR 279,396 is a paromomycin-based topical cream that has shown some suggestion of being effective for the treatment of non-serious, non-complicated cutaneous leishmaniasis in previous clinical studies. The goal of this study is to expand those observations in a larger, more rigorous study to clearly define the efficacy of this product and collect information about adverse effects. Subjects will be randomized to receive either WR 279,396 or vehicle placebo; applied twice a day for 20 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-75 years
* Lesions must measure at least 1 cm and be primarily ulcerative
* Have cutaneous leishmaniasis proven parasitologically in the lesion selected for study
* Must have given written informed consent to participate in the study

Exclusion Criteria:

* Known drug intolerance to aminoglycosides in the patient or immediate family
* Previous use of antileishmanial drugs (within 3 months) or present use of routinely nephrotoxic or ototoxic drugs
* Patients with tuberculosis under treatment
* Potential for follow-up: have less than 7 months time remaining in present address and/or plan to leave the area for more than 30 days
* Extent of disease: more than 5 lesions or lesion equal to or greater than 5 cm or a lesion less than 5 cm from the eye, or a lesion in the face that, in the opinion of the attending dermatologist could potentially cause significant disfigurement
* Location of disease: mucosal involvement
* Disseminated disease: clinically significant lymphadenitis with nodules that are painful and greater than 1 cm in size in the lymphatic drainage of the ulcer
* Concomitant medical problems: significant medical problems of the kidney or liver as determined by history and by the following laboratory studies:
* Hearing abnormality
* Ongoing pregnancy or have plans to become pregnant
* Females of child bearing age (Tunisia Only)
* Signs or symptoms of peripheral neuropathy

Kidney: clinically significant abnormalities of urine analysis, serum levels of creatinine, BUN, total proteins greater than the upper limit of normal for the laboratory.

Liver: AST or ALT greater than the upper limit of normal for the laboratory General: glucose, Na+, or K+ greater than the upper limit of normal for the laboratory

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2003-03; Primary Completion 2004-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afif Ben Salah, M.D., Ph.D., Principal Investigator — Institute Pasteur Tunisia
Locations (2):
- Medical Center Institut Pasteur, Paris, France
- Institue Pasteur, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with WRAIR

REFERENCES:
- [Result] Ben Salah A, Buffet PA, Morizot G, Ben Massoud N, Zaatour A, Ben Alaya N, Haj Hamida NB, El Ahmadi Z, Downs MT, Smith PL, Dellagi K, Grogl M. WR279,396, a third generation aminoglycoside ointment for the treatment of Leishmania major cutaneous leishmaniasis: a phase 2, randomized, double blind, placebo controlled study. PLoS Negl Trop Dis. 2009;3(5):e432. doi: 10.1371/journal.pntd.0000432. Epub 2009 May 5. PMID 19415122

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WR 279,396 | Placebo
Started | 50 | 42
Completed | 49 | 41
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WR 279,396 | Placebo | Total
Number analyzed (Participants) | 50 | 42 | 92
Age, Customized [Number; unit: years]
  <18 years | 47 | 33 | 80
  >18 years | 3 | 9 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 15 | 38
  Male | 27 | 27 | 54
Region of Enrollment [Number; unit: participants]
  France | 5 | 5 | 10
  Tunisia | 45 | 37 | 82

OUTCOME MEASURES:

1. Primary Outcome: Complete Clinical Response (CCR) of Lesion at Days 50, 100 and 180 (+7 Days)
Description: CCR is defined as at least 50% reduction, from baseline, in index lesion area of ulceration at study days 50, 100 and 180 (+ 7 days). Randomized subjects were compared using the uncorrected Fisher's exact test. Confidence intervals (95%) were constructed on the difference between the two group proportions. The log-rank test was used to compare the time to complete re-epithelialization of the index lesion without relapse. Cure of all subjects lesions was also compared using the Fisher's exact test. To adjust for baseline differences in the treatment groups, a linear model for the proportion of subjects achieving CCR was fit for each baseline variable of interest with covariates for treatment group and the baseline variable. The Breslow-Day test was used to examine whether the effect of WR 279,396 varied between subgroups
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | WR 279,396 | Placebo
Number analyzed (Participants) | 50 | 42
Participants
  CCR | 47 | 30
  CCR Failure | 3 | 12

2. Primary Outcome: Safety of WR 279,396 (AEs and SAEs)
Description: Safety was evaluated on each day during daily administration of the topical products. Subjects were observed and questioned for the occurrence of solicited local side effects (eg, pain, erythema, edema) and solicited systemic side effects (eg, vertigo, tinnitus, diminished hearing). Non-solicited AE evaluations included spontaneous reports from subjects and clinical observations.
Time Frame: 180 days
Population: All solicited local and systemic AEs and SAEs including immediate and delayed reactions that occurred during this study are summarized.
Measure: Number; unit: Adverse Events
Arm/Group | WR 279,396 | Placebo
Number analyzed (Participants) | 50 | 42
Adverse Events
  Solicated AEs- Mild | 49 | 40
  Solicited AEs- Moderate | 11 | 5
  Solicited AEs- Severe | 2 | 2
  Non-Solicited AEs- Mild | 13 | 20
  Non-Solicited AEs- Moderate | 10 | 10
  Non-Soliciated AEs- Severe | 0 | 0
  SAEs | 1 | 0

3. Secondary Outcome: Time to Complete Re-epithelialization of the Index Lesion Ulcer Without Relapse
Description: 100% re-epithelialization of the index lesion without having had a relapse. The log-rank test was used to compare the time to complete re-epithelialization.
Time Frame: 180 days
Population: Days to 100% re-epithelialization of index lesion. Volunteer Identification Number (VIN). VINs 17, 72, and 109 failed to meet 100% re-epithelialization
Measure: Count of Participants; unit: Participants
Groups:
- Day 20: 100% Re-epithelialization by day 20
- Day 50: 100% Re-epithelialization by day 50
- Day 100: 100% Re-epithelialization by day 100
- Day 180 (+7 Days): 100% Re-epithelialization by day 180 (+7 days)
Arm/Group | Day 20 | Day 50 | Day 100 | Day 180 (+7 Days)
Number analyzed (Participants) | 92 | 92 | 92 | 92
Participants
  WR 279,396: number analyzed (Participants) | 50 | 50 | 50 | 50
  WR 279,396 | 10 | 34 | 4 | 1
  Placebo: number analyzed (Participants) | 42 | 42 | 42 | 42
  Placebo | 20 | 10 | 9 | 1

4. Secondary Outcome: Final Cure Rate by Subject of All Lesions
Description: Final cure rate by subject was determined using the Fisher's exact test. To adjust for baseline differences in the treatment groups, a linear model for the proportion of subjects achieving CCR was fit for each baseline variable of interest with covariates for treatment group and the baseline variable.
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | WR 279,396 | Placebo
Number analyzed (Participants) | 50 | 42
Participants
  CCR | 46 | 29
  Treatment Failure | 4 | 13

5. Secondary Outcome: Rate of Relapse
Description: Relapse is defined as enlargement of the index lesion compared to previous measurement at any time after day 50 (+ 7 days) or not demonstrating CCR by study day 180. CCR was compared using uncorrected Fisher's exact test.
  Confidence intervals (95%) were constructed on the difference between the two group proportions. The log-rank test was used to compare the time to complete re-epithelialization of the index lesion without relapse. Cure of all subjects lesions was also compared using the Fisher's exact test. To adjust for baseline differences in the treatment groups, a linear model for the proportion of subjects achieving CCR was fit for each baseline variable of interest with covariates for treatment group and the baseline variable.
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | WR 279,396 | Placebo
Number analyzed (Participants) | 50 | 42
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: Duration of study (180 days (+7 days)
Description: AEs were evaluated on each day during daily administration of the topical products. Subjects were observed and questioned for the occurrence of solicited local side effects (eg, pain, erythema, edema) and solicited systemic side effects (eg, vertigo, tinnitus, diminished hearing). Non-solicited AE evaluations included spontaneous reports from subjects and clinical observations.
  * Immediate: observed within 30 minutes of application
  * Delayed: observed just prior to next application
Arm/Group | WR 279,396 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/42
Other Adverse Events (participants affected / at risk) | 16/50 | 12/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WR 279,396 (N=50) | Placebo (N=42)
Arm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WR 279,396 (N=50) | Placebo (N=42)
Immediate - Local pain (General disorders) | 7 (7) | 6 (6) — Mild
Immediate - Local pain (General disorders) | 0 (0) | 0 (0) — Moderate
Immediate - Local pain (General disorders) | 0 (0) | 0 (0) — Severe
Immediate - Local Erythema (Skin and subcutaneous tissue disorders) | 15 (15) | 10 (10) — Mild
Immediate - Local Erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) — Moderate
Immediate - Local Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Severe
Immediate - Local Edema (Metabolism and nutrition disorders) | 1 (1) | 2 (2) — Mild
Immediate - Local Edema (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Moderate
Immediate - Local Edema (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Severe
Immediate - Vertigo (Nervous system disorders) | 0 (0) | 1 (1)
Immediate - Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Immediate - Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0)
Delayed - Local Pain (General disorders) | 9 (9) | 5 (5) — Mild
Delayed - Local Pain (General disorders) | 0 (0) | 0 (0) — Moderate
Delayed - Local Pain (General disorders) | 0 (0) | 0 (0) — Severe
Delayed - Local Erythema (Skin and subcutaneous tissue disorders) | 15 (15) | 10 (10) — Mild
Delayed - Local Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) — Moderate
Delayed - Local Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Severe
Delayed - Local Edema (Metabolism and nutrition disorders) | 1 (1) | 3 (3) — Mild
Delayed - Local Edema (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Moderate
Delayed - Local Edema (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Severe
Delayed - Vertigo (Nervous system disorders) | 0 (0) | 3 (3)
Delayed - Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0)
Delayed - Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) — Moderate
Application site erythema (General disorders) | 1 (1) | 1 (1) — Moderate
Application site erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Mild
Application site oedema (Metabolism and nutrition disorders) | 1 (1) | 2 (2) — Mild
Fatigue (General disorders) | 1 (1) | 1 (1) — Mild
Fatigue (General disorders) | 0 (0) | 1 (1) — Moderate
Nodule (General disorders) | 1 (1) | 0 (0) — Mild
Pain (General disorders) | 1 (1) | 4 (4) — Mild
Pain (General disorders) | 2 (2) | 0 (0) — Moderate
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) — Moderate
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) — Mild
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Severe
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Mild
Headache (Nervous system disorders) | 1 (1) | 1 (1) — Mild
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Moderate
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) — Mild
Dermatitis contact (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4) — Mild
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) — Moderate
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Moderate
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Mild
Eye pain (Eye disorders) | 0 (0) | 1 (1) — Mild
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Mild
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Mild
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Mild
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) — Moderate
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) — Mild
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) — Mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No